CLINICAL TRIAL: NCT04459234
Title: KETACANCER: Prospective Multicentre Study of the Use of Ketamine in the Treatment of Refractory Chronic Pain in the French CLCC
Brief Title: Prospective Multicentre Study of the Use of Ketamine in the Treatment of Refractory Chronic Pain in the French CLCC
Acronym: KETACANCER
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET20-130 - KETACANCER
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Cancer; Chronic Pain; Neuropathic Pain; Opioid Use
Keywords: Cancer; Palliative care; Ketamine; Chronic pain
MeSH Terms: conditions — Neoplasms; Chronic Pain; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ketamine use in CLCC sites (indication and administration protocol) — Collection of information concerning Ketamine use by French CLCCs pain teams (first prescription):
  1. Indications : analgesic treatment of cancer chronic pain, analgesic treatment for a post-cancer treatment chronic pain, help for withdrawal from opioid treatment prescribed for a chronic cancer pain
  2. Administration protocol: route, posology, duration, administration sequence, premedication
  3. Antalgic efficacy
  4. Tolerance profile
  5. Quality of life, anxiety and depression evaluations

SUMMARY:
The primary objective of this study is to describe the administration practices of the antalgic Ketamine in French CLCC (Centre de Lutte Contre le Cancer) in terms of indication (neuropathic sequelae pains, morphine additional effect or morphine withdrawal, intensity, localisation…) and administration protocol (route, posology, duration, administration sequence, premedication).

The secondary objectives are to evaluate in the context of cancer, the analgesic efficacy, the tolerance profile (biological and clinical toxicities) and the quality of life, including anxiety and depression.

In addition, the described parameters will be evaluated as safety and efficacy predictive factors of the Ketamine in oncology.

DETAILED DESCRIPTION:
Almost 382,000 new cancers have been diagnosed in France in 2018. Regular progresses in their management have improved the overall survival of patients, sometimes with sequelae that may be particularly painful. Thus for 20 to 45% of patients treated for breast cancer, pain persists 5 years later.

If remission is a regularly reached target, cancer was also the cause of 157,000 deaths in 2018 in France, preceded by months or years of progression of a chronic disease that regularly causes pain. Pain during cancer (chronic cancer pain for CIM-11) remains a frequent symptom, and its prevalence has slightly changed during the last 20 years.

In the European EPIC study, carried out in 2006, 76% of the cancer patients (and 62% of French patients) presented moderate to severe pains linked to cancer, daily for more than half of them.

Even when identified, chronic cancer pain is still under-treated in 25 to 60% of cases worldwide, including in the most developed countries.

When well-managed, pain's management now allows the relief of almost 80% of patients. Pain's management is based in particular on a precise and adapted use of the different opioids through different routes of administration (oral, transdermal, trans-mucosal, parenteral, etc.).

A neuropathic component of pain exists in almost a third of cases and may require specific treatments when opioids are insufficient. In all cases, the treatment is integrated into a multidisciplinary management, in connection with the ongoing oncological treatments, the loco-regional treatments available (radiotherapy, interventional radiology, etc.) and with an adapted psychosocial management.

Ketamine is an NMDA receptor antagonist (N-Methyl-D-Aspartate) indicated as a high dose anesthetic. It is used in the context of peri-operative pain for its anti-hyperalgesic properties. These properties have led to its use also in palliative care (outside the marketing authorization [AMM]) to treat hyperalgesia linked to the use of high-doses of opioids, as well as depression. For non-cancer pains, ketamine is widely used by centres and consultations specialized in refractory chronic pain management in different pains not relieved by standard treatments: neuropathic pain, fibromyalgia, etc., or even in opioids weaning aid.

The bibliographic data are not homogeneous and of low quality. Despite the weakness of the available data, ketamine is widely used in France in chronic pain in situation of therapeutic impasse. The protocols used vary according to the prescribers and services practices: venous route in general, sometimes subcutaneous or even oral; doses varying from 30 to 200 mg / day, infusion duration varying from a few hours to several days, discontinuous administration by cycle or continuous administration, etc.

Current knowledge is too limited in oncology to have a consensus on the use of ketamine :

* Often retrospective studies with heterogeneous treatment protocols;
* Studied populations also heterogeneous, with insufficiently documented indications;
* Staff not able to answer adequately the questions raised. This situation largely explains the heterogeneity of the Ketamine practices of use in oncology

It is essential to draw up an inventory of the ketamine use by the French CLCCs pain teams and to identify the profile of patients in whom i) the treatment is ineffective and must be avoided regarding toxicities ii) the potential efficacy required further investigations. Built on a methodology close to the OKAPI study, the KETACANCER study will enable to compare indirectly the results of the two studies.

To do this, it is proposed to conduct the KETACANCER prospective study in a precise population defined a priori, and corresponding to the following indications:

* Neuropathic sequelae pain
* Additional effect of morphine
* Morphine weaning.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old at the day of consenting to the study
* Patient followed for a solid tumour or a hematological malignancy (treated or under treatment)
* Patient presenting cancer chronic pain or post cancer treatment pain
* Patient followed by a CLCC's intractable chronic pain consultation or centre
* Patient with an indication of 1st Ketamine course:
* Analgesic treatment of cancer chronic pain
* Analgesic treatment for a post-cancer treatment chronic pain
* Help for withdrawal from opioid treatment prescribed for a chronic cancer pain
* Patient not previously treated by Ketamine
* Patient covered by a medical insurance
* Patient and/or family did not decline data collection after complete information (information sheet)

Exclusion Criteria:

* Patient presenting chronic pains not related to cancer or its treatments
* Patient with a proven psychotic history
* Patient who is not fluent enough in French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, multicentre study, considered as " non-RIPH (Recherche n'Impliquant pas la Personne Humaine ". Indeed, the patient's participation in the study and the completion of the various questionnaires has no impact on patient's safety and is not likely to change his/her management. The treatment will be conducted according to the standard practices of each participating site (continuous or discontinuous protocol, dosage, rhythm of administration, monitoring, etc.). The questionnaires and scales used in this study are part of the recommended tools for monitoring this population.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Describe the administration practices of the antalgic Ketamine in French CLCC (Centre de Lutte Contre le Cancer) in terms of indication | Up to 3 months after inclusion
  neuropathic sequelae pains, morphine additional effect or morphine withdrawal, intensity, localisation
Describe the administration practices of the antalgic Ketamine in French CLCC (Centre de Lutte Contre le Cancer) in terms of administration protocol | Up to 3 months after inclusion
  route, posology, duration, administration sequence, premedication

SECONDARY OUTCOMES:
Evaluate in the context of cancer the antalgic efficacy | Up to 3 months after inclusion
  Questionnaire: NPSI
Evaluate in the context of cancer the antalgic efficacy | Up to 3 months after inclusion
  Questionnaire: DN4
Evaluate in the context of cancer the antalgic efficacy | Up to 3 months after inclusion
  Questionnaire: PGIC
Evaluate in the context of cancer the tolerance profile | Up to 3 months after inclusion
  The safety will be described mainly on the frequency of adverse events coded using the common toxicity criteria (NCI-CTCAE v5.0) grade. Descriptive statistics will be provided for characterizing and assessing patient's tolerance to treatment. Adverse events will be coded according to the MedDRA®.
Evaluate in the context of cancer the quality of life including anxiety and depression | Up to 3 months after inclusion
  Numeric scale (from 0 : no pain to 10: maximum pain)
Evaluate in the context of cancer the quality of life including anxiety and depression | Up to 3 months after inclusion
  Questionnaire: HADS

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle CHVETZOFF, MD, Principal Investigator — Centre Leon Berard
Locations (12):
- France (12):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancérologie de Montpellier, Montpellier
  - Institut Curie, Paris
  - Institut Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Institut Universitaire du Cancer (IUCT), Toulouse
  - Institut de Cancérologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif